CLINICAL TRIAL: NCT04235699
Title: Benefits of Ketogenic Diet in Patients With Heart Failure With Preserved Ejection Fraction: A Pilot Study
Brief Title: Ketogenic Diet in Patients With Heart Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped recruiting during the pandemic and then PI left OSU.
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019H0255
Record Dates: First submitted 2020-01-15; First posted 2020-01-22 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic Diet (Experimental): This arm will be provided food to induce a state of nutritional ketosis in each person as defined as blood [3-OHB] ≥0.5 mM.
  Interventions: Other: Nutritional and Dietary Manipulation
- Low-fat mixed Diet (Experimental): This arm will be provided food consisting of ~25% fat, and the remaining calories from carbohydrate (~55% after accounting for protein at ~20%).
  Interventions: Other: Nutritional and Dietary Manipulation

INTERVENTIONS:
Other: Nutritional and Dietary Manipulation — Participants will undertake a controlled feeding intervention. All food will be prepared and delivered to participants by research staff. Participants will be asked to exclusively eat what is provided to them in efforts to control any dietary effects.

SUMMARY:
This study is being done to evaluate the effects of a low carbohydrate ketogenic diet on exercise tolerance in patients with Heart Failure with Preserved Ejection Fraction (HFpEF), also known as Diastolic Heart Failure (DHF).

DETAILED DESCRIPTION:
Patients will be randomized to either a ketogenic diet, or a low-fat diet higher in carbohydrate and based on current dietary guidelines. Regardless of what group you are randomized to, you will consume the diet for a period of 4 weeks. All foods will be prepared by our research group and provided to you. Both diets will be based on an approximately 25% reduction in your dietary caloric requirements, so some weight loss may occur over the 4-week intervention.

Primary data collection will occur at baseline and at four weeks, with more frequent monitoring of blood markers, blood pressure, heart rate, and overall health. Throughout the duration of the study, you will be continued on standard heart failure therapies as guided by your treating physician. The duration of the study is expected to last for approximately 6 weeks. This includes all before and after testing, as well as the 4 weeks on diet.

All patients will undergo a resting MRI scan of the heart at enrollment (baseline), and again at the end of the 4-week diet. You will not receive any injections.

All participants will also undergo a cardiopulmonary stress test (CPET, also known as VO2 testing) at enrollment (baseline) and again at the end of the 4-week dietary intervention. During the Cardiopulmonary stress testing you will be asked to exercise on a treadmill while breathing into a mask.

All participants will also undergo body fat and body fluid composition by dual-energy X-ray absorptiometry (DXA) at enrollment (baseline) and again at the end of the 4 week dietary intervention. You will be exposed to a very small amount of radiation by the DXA scanner used to measure your body composition. However, amount of radiation used in DXA is extremely low (by comparison, a standard chest x-ray is 125 times more radiation than a DXA scan).

Blood tests will be performed at enrollment (baseline) and again at the end of the 4 week dietary intervention. Blood draws may cause discomfort at the skin puncture site and a small bruise may develop that may persist for several weeks. There is also a small possibility of an infection. These risks are identical to standard clinical blood draws.

After 2-weeks, and again after 4 weeks on diet, all participants will undergo a clinical examination by a cardiologist.

All participants will be provided with a handheld glucometer and test strips to check ketone levels daily in the morning after an overnight fast. This requires a finger prick to obtain the drop of blood required for the test. The finger stick may cause a slight immediate discomfort at the specific stick site. Subjects will also be required to check and record ketones 4x/day on one day per week to capture a more accurate record of ketone levels during waking hours. You will bring the glucometer readings with you when you pick up food so that the results can be downloaded and recorded by a member of the research team.

Patients on either diet will personally pick up food 3X per week. Patients will weigh-in and have their heart rate and blood pressure checked at the time of each food pick up. The MRI, the cardiopulmonary stress test and all blood testing will be done at the Ross Heart Hospital or the Davis Heart and Lung Research Institute. The DXA testing, as well as the food pickup will be done at the Physical Activity and Educational Services (PAES) building on The Ohio State University campus.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old and ≤ 75 years old & willingness to be randomized to either diet
* Confirmed diagnosis of heart failure with ejection fraction ≥50% (NYHA Class II-IV)
* On optimal medical therapy for at least 3 months as determined by the treating physician
* Body Mass Index (BMI) ≥ 25
* Ability to participate in exercise treadmill testing

Exclusion Criteria:

* Contraindications to MRI including pregnancy
* Diagnosis of diabetes mellitus treated with insulin or SGLT2 inhibitors.
* History of diabetic ketoacidosis
* Recent (within 30 days) or planned (within 30 days) cardiac revascularization
* Recent acute myocardial infarction or acute coronary syndrome (30 days)
* Body Mass Index (BMI) < 25, or BMI > 40
* Hepatic cirrhosis
* Use of metformin > 1700 mg daily
* Left ventricular ejection fractions < 50%
* Prior diagnosis of moderate to severe COPD
* Uncontrolled systemic systolic/diastolic hypertension (SBP > 150 mmHg or DBP > 90 mmHg)
* Echocardiographic evidence of significant valvular disease
* History of ventricular tachycardia or SCD
* Untreated moderate or severe sleep apnea

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-12-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in maximal exercise performance | Baseline and end of study participation, 6 weeks
  Participants will undergo VO2 max testing, conducted by trained professionals. VO2 max testing analyses will determine changes in maximal exercise performance

SECONDARY OUTCOMES:
Change in CMR measures of cardiac function | Baseline and end of study participation, 6 weeks
  Participants will undergo MRI scans, conducted by trained professionals. MRI imaging analyses will determine cardiac function. The images will be analyzed by trained imaging professionals to determine overall change in cardiac function.
Change in NYHA class | Baseline and end of study participation, 6 weeks
  NYHA class will be determined by clinical examination by a qualified cardiovascular physician
Change in Quality of Life Questionnaire | Baseline and end of study participation, 6 weeks
  Participants will complete a quality of life questionnaire several times throughout the study. The questions are divided into three areas: Dyspnea, Fatigue and Emotional Function. The scores for each area are added up and divided by the number of questions. A 7-point scale is used for all areas where 1 is the best and 7 is the worst.
Change in Serologic Markers | Baseline and end of study participation, 6 weeks
  Cardio-metabolic risk markers will be determined through blood samples taken throughout the study. We will look at B-natriuretic peptide (BNP), total cholesterol, HDL, LDL, triglycerides, lipoprotein particle distribution, fasting blood glucose, serum potassium, sodium, and magnesium.

CONTACTS AND LOCATIONS:
Overall Officials: Sitaramesh Emani, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Final results will be published via peer-review process.
Supporting Information: Study Protocol, ICF